CLINICAL TRIAL: NCT01973231
Title: Efficacy and Safety of Liraglutide Versus Lixisenatide as add-on to Metformin in Subjects With Type 2 Diabetes
Acronym: LIRA-LIXI™
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-3867; 2012-004984-27 (EudraCT Number); U1111-1136-3644 (Other: WHO)
Record Dates: First submitted 2013-10-23; First posted 2013-10-31 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; lixisenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin + liraglutide 1.8 mg (Experimental)
  Interventions: Drug: liraglutide
- Metformin + lixisenatide 20 microg (Active Comparator)
  Interventions: Drug: lixisenatide

INTERVENTIONS:
Drug: liraglutide — Starting dose of 0.6 mg/day, with weekly dose escalations of 0.6 mg/day until the maintenance dose of 1.8 mg/day is reached. Administered s.c. (subcutaneously, under the skin) once daily in addition to the subject's stable pre-trial metformin (equal to or above 1000 mg/day and up to 3000 mg/day).
  Arms: Metformin + liraglutide 1.8 mg
Drug: lixisenatide — Starting dose of 10 microg to be administered s.c. once daily, within the hour prior to the first meal of the day or the evening meal in addition to subject's stable pre-trial metformin (equal to or above 1000mg/day and up to 3000mg/day). Dose escalation to 20 microg s.c. once daily from day 15 after randomization.
  Arms: Metformin + lixisenatide 20 microg

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the efficacy and safety of liraglutide versus lixisenatide as add-on to metformin in subjects with type 2 diabetes (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Subjects diagnosed with T2DM and on unchanged metformin treatment at the maximum tolerated dose (at least 1000 mg/day and up to 3000 mg/day) for at least 90 days prior to screening
* HbA1c 7.5 - 10.5% (53 mmol/mol - 91 mmol/mol) (both inclusive)
* Body Mass Index (BMI) equal to or above 20 kg/m^2

Exclusion Criteria:

* Female of child-bearing potential who is pregnant, breast-feeding or intend to become pregnant or is not using adequate contraceptive methods. (Adequate contraceptive measures as required by local law or practice)
* Treatment with glucose lowering agent(s) other than stated in the inclusion criteria in a period of 90 days prior to screening. Exception is short-term treatment (equal to or below 7 days in total) with insulin in connection with intercurrent illness
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Screening calcitonin value equal to or above 50 ng/L
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2)
* Impaired liver function, defined as alanine aminotransferase (ALAT) equal to or above 2.5 times upper normal limit (UNL)
* Impaired renal function defined as estimated glomerular filtration rate (eGFR) below 60 mL/min/1.73 m^2 per Modification of Diet in Renal Disease (MDRD) formula
* Any episode of unstable angina, acute coronary event, cerebral stroke/transient ischemic attack (TIA) or other significant cardiovascular event as judged by the investigator within 90 days prior to screening
* Heart failure, New York Heart Association (NYHA) class IV
* Uncontrolled hypertension (defined as systolic blood pressure equal to or above 180 mmHg and/or diastolic blood pressure equal to or above 100 mmHg)
* Diagnosis of malignant neoplasm in the previous 5 years (except basal cell skin cancer or squamous cell skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (55):
- Czechia (5):
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Mladá Boleslav
  - Novo Nordisk Investigational Site, Olomouc
  - Novo Nordisk Investigational Site, Pilsen
  - Novo Nordisk Investigational Site, Prostějov
- Finland (5):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Jyväskylä
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Pori
  - Novo Nordisk Investigational Site, Rovaniemi
- France (7):
  - Novo Nordisk Investigational Site, Boulogne-Billancourt
  - Novo Nordisk Investigational Site, Corbeil-Essonnes
  - Novo Nordisk Investigational Site, Hinx
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Saint-Herblain
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (9):
  - Novo Nordisk Investigational Site, Bad Lauterberg im Harz
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Bochum
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Lampertheim
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Saint Ingbert
- Hungary (6):
  - Novo Nordisk Investigational Site, Baja
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Gyula
  - Novo Nordisk Investigational Site, Pécs
  - Novo Nordisk Investigational Site, Salgótarján
  - Novo Nordisk Investigational Site, Szeged
- Italy (5):
  - Novo Nordisk Investigational Site, Catania
  - Novo Nordisk Investigational Site, Cittadella (PD)
  - Novo Nordisk Investigational Site, Padua
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Terni
- Latvia (2):
  - Novo Nordisk Investigational Site, Ogre
  - Novo Nordisk Investigational Site, Riga
- Lithuania (4):
  - Novo Nordisk Investigational Site, Kaunas
  - Novo Nordisk Investigational Site, Klaipėda
  - Novo Nordisk Investigational Site, Šiauliai
  - Novo Nordisk Investigational Site, Vilnius
- United Kingdom (12):
  - Novo Nordisk Investigational Site, Basingstoke
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Chester
  - Novo Nordisk Investigational Site, Chiswick
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Derby
  - Novo Nordisk Investigational Site, Devon
  - Novo Nordisk Investigational Site, Great Yarmouth
  - Novo Nordisk Investigational Site, Lancaster
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Sandbach
  - Novo Nordisk Investigational Site, Taunton

REFERENCES:
- [Result] Nauck M, Rizzo M, Johnson A, Bosch-Traberg H, Madsen J, Cariou B. Once-Daily Liraglutide Versus Lixisenatide as Add-on to Metformin in Type 2 Diabetes: A 26-Week Randomized Controlled Clinical Trial. Diabetes Care. 2016 Sep;39(9):1501-9. doi: 10.2337/dc15-2479. Epub 2016 Jun 16. PMID 27311491
- [Derived] Hunt B, Vega-Hernandez G, Valentine WJ, Kragh N. Evaluation of the long-term cost-effectiveness of liraglutide vs lixisenatide for treatment of type 2 diabetes mellitus in the UK setting. Diabetes Obes Metab. 2017 Jun;19(6):842-849. doi: 10.1111/dom.12890. Epub 2017 Feb 23. PMID 28124820
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 56 sites in 9 countries; Czech Republic (5), Finland (4), France (6), Germany (8), Hungary (6), Italy (5), Latvia (6), Lithuania (5) and UK (11).
Groups:
- Liraglutide: Liraglutide was administered subcutaneously (s.c.; under the skin) once daily in addition to the subject's stable pre-trial metformin (maximum tolerated dose, equal to or above 1000 mg/day and up to 3000 mg/day) for a total duration of 26 weeks. Starting dose of liraglutide was 0.6 mg/day, with weekly dose escalations of 0.6 mg/day until the maintenance dose of 1.8 mg/day was reached.
- Lixisenatide: Lixisenatide was administered s.c. once daily, within the hour prior to the first meal of the day or the evening meal in addition to subject's stable pre-trial metformin (maximum tolerated dose, equal to or above 1000mg/day and up to 3000mg/day) for a total duration of 26 weeks. Starting dose of lixisenatide was 10 µg once daily, the dose was escalated to 20 µg once daily from day 15 after randomisation.
Period: Overall Study
Arm/Group | Liraglutide | Lixisenatide
Started | 202 | 202
Completed | 191 | 190
Not Completed | 11 | 12
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — unclassified | 2 | 1
Not completed — Withdrawal by Subject | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Lixisenatide | Total
Number analyzed (Participants) | 202 | 202 | 404
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (10.6) | 56.1 (10.0) | 56.2 (10.3)
Gender [Count of Participants; unit: Participants]
  Female | 70 | 90 | 160
  Male | 132 | 112 | 244
Glycosylated Haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin] | 8.40 (0.723) | 8.43 (0.785) | 8.41 (0.754)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 10.47 (2.368) | 10.25 (2.254) | 10.36 (2.312)
Body Weight [Mean (Standard Deviation); unit: kg] | 101.89 (23.344) | 100.58 (19.949) | 101.24 (21.696)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c) From Baseline
Description: Change from baseline in HbA1c after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: The full analysis set (FAS) included all randomised subjects. Missing values were imputed using predicted values from the mixed model for repeated measurements (MMRM) model. Due to missing HbA1c post baseline data, 194 and 191 subjects in liraglutide and lixisenatide treatment group, respectively were included in the HbA1c analysis.
Measure: Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin
Arm/Group | Liraglutide | Lixisenatide
Number analyzed (Participants) | 194 | 191
Percent (%) glycosylated haemoglobin | -1.809 (0.9159) | -1.238 (1.0085)

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline
Description: Change from baseline in FPG after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects. Missing values were imputed using predicted values from the MMRM model. Due to missing FPG post baseline data, 194 and 189 subjects in liraglutide and lixisenatide treatment group, respectively were included in the FPG analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide | Lixisenatide
Number analyzed (Participants) | 194 | 189
mmol/L | -2.904 (2.2309) | -1.644 (2.1511)

3. Secondary Outcome: Change in Body Weight From Baseline
Description: Change from baseline in body weight after 26 weeks of treatment.
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects. Missing values were imputed using predicted values from the MMRM model. Due to missing body weight post baseline data, 194 and 191 subjects in liraglutide and lixisenatide treatment group, respectively were included in the body weight analysis.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide | Lixisenatide
Number analyzed (Participants) | 194 | 191
kg | -4.24 (4.273) | -3.69 (4.746)

4. Secondary Outcome: Subjects Who Achieve HbA1c Below 7.0% (53 mmol/Mol) (American Diabetes Association (ADA) Target) (Yes/no)
Description: Subjects who achieved HbA1c below 7.0% (53 mmol/mol) after 26 weeks of treatment (yes/no).
Time Frame: After 26 weeks of treatment
Population: The FAS included all randomised subjects. Missing values were imputed using predicted values from the MMRM model. Due to missing HbA1c post baseline data, 194 and 191 subjects in liraglutide and lixisenatide treatment group, respectively were included in the HbA1c analysis.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Liraglutide | Lixisenatide
Number analyzed (Participants) | 194 | 191
percentage (%) of subjects
  Yes | 74.2 | 45.5
  No | 25.8 | 54.5

5. Secondary Outcome: Subjects Who Achieve HbA1c Equal to or Below 6.5% (48 mmol/Mol) (American Association of Clinical Endocrinologists [AACE] Target) (Yes/no)
Description: Subjects who achieved HbA1c below equal to or below 6.5% (48 mmol/mol) after 26 weeks of treatment (yes/no).
Time Frame: After 26 weeks of treatment
Population: as for outcome 4
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Liraglutide | Lixisenatide
Number analyzed (Participants) | 194 | 191
percentage (%) of subjects
  Yes | 54.6 | 26.2
  No | 45.4 | 73.8

6. Secondary Outcome: Subjects Who Achieve HbA1c Below 7.0% (53 mmol/Mol) and no Weight Gain (Yes/no)
Description: Subjects who achieved HbA1c below 7.0% (53 mmol/mol) and no weight gain after 26 weeks of treatment (yes/no).
Time Frame: After 26 weeks of treatment
Population: The FAS included all randomised subjects. Missing values were imputed using predicted values from the MMRM model. Due to missing HbA1c post-baseline data, 194 and 191 subjects in liraglutide and lixisenatide treatment group, respectively were included in the HbA1c analysis.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Liraglutide | Lixisenatide
Number analyzed (Participants) | 194 | 191
percentage (%) of subjects
  Yes | 66.5 | 41.9
  No | 33.5 | 58.1

7. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: A Treatment Emergent Adverse Event (TEAE) was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment. Severity was assessed by investigator.
Time Frame: Weeks 0-26
Population: The safety analysis set (SAS) included all subjects who received at least one dose of any of the trial products.
Measure: Number; unit: events
Arm/Group | Liraglutide | Lixisenatide
Number analyzed (Participants) | 202 | 202
events
  Events | 540 | 435
  Serious | 13 | 7
  Severe | 10 | 3
  Moderate | 109 | 84
  Mild | 421 | 348

ADVERSE EVENTS:
Time Frame: Weeks 0-26
Description: The SAS included all subjects who received at least one dose of any of the trial products.
Arm/Group | Liraglutide | Lixisenatide
Serious Adverse Events (participants affected / at risk) | 12/202 | 7/202
Other Adverse Events (participants affected / at risk) | 90/202 | 83/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=202) | Lixisenatide (N=202)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) — Complete preferred term of the AE: Anxiety disorder due to a general medical condition
Prostatic dysplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=202) | Lixisenatide (N=202)
Diarrhoea (Gastrointestinal disorders) | 25 (39) | 20 (22)
Dyspepsia (Gastrointestinal disorders) | 11 (11) | 6 (9)
Nausea (Gastrointestinal disorders) | 44 (67) | 44 (60)
Vomiting (Gastrointestinal disorders) | 14 (18) | 18 (22)
Nasopharyngitis (Infections and infestations) | 13 (13) | 20 (22)
Lipase increased (Investigations) | 17 (17) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 13 (13) | 5 (5)
Headache (Nervous system disorders) | 15 (31) | 17 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of plans by any investigator to publish and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager before submission for comments. Comments will be given within four weeks from receipt of the planned communication.